CLINICAL TRIAL: NCT00579020
Title: An Evaluation of Moxidex Ophthalmic Solution for Treatment of Marginal Corneal Infiltrates
Brief Title: A Phase II Study of Moxidex Ophthalmic Solution for Treatment of Marginal Corneal Infiltrates
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-05-04
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Corneal Infiltrates
Keywords: cornea; inflammation; blepharitis; lid infection
MeSH Terms: conditions — Corneal Diseases; Inflammation; Blepharitis | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moxidex (Experimental): Moxifloxacin/dexamethasone phosphate ophthalmic solution, one drop in cul-de-sac and 4 drops on closed lids of study eye(s), four times a day, for seven days
  Interventions: Drug: Moxifloxacin/dexamethasone phosphate ophthalmic solution
- Moxifloxacin (Active Comparator): Moxifloxacin ophthalmic solution 0.5%, one drop in cul-de-sac and 4 drops on closed lids of study eye(s), four times a day, for seven days
  Interventions: Drug: Moxifloxacin ophthalmic solution 0.5%
- Dexamethasone (Active Comparator): Dexamethasone phosphate solution, 0.1%, one drop in cul-de-sac and 4 drops on closed lids of study eye(s), four times a day, for seven days
  Interventions: Drug: Dexamethasone phosphate solution, 0.1%

INTERVENTIONS:
Drug: Moxifloxacin/dexamethasone phosphate ophthalmic solution
  Other Names: Moxidex
  Arms: Moxidex
Drug: Moxifloxacin ophthalmic solution 0.5%
  Arms: Moxifloxacin
Drug: Dexamethasone phosphate solution, 0.1%
  Arms: Dexamethasone

SUMMARY:
The purpose of the study is to determine whether Moxidex ophthalmic solution is safe and effective in treating marginal corneal infiltrates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of marginal corneal infiltrates of size equal to or less than 1.5mm in diameter, with mild, moderate or severe bulbar conjunctival injection in at least one eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Age related.
* Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with resolution of all corneal stromal infiltrate(s) in study eye at Test of Cure (TOC) Visit (Day 10) | Day 10

SECONDARY OUTCOMES:
Percentage of patients with eradication of pre-therapy pathogens from the lid of the study eye at TOC Visit (Day 10) | Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937, Fort Worth, Texas, United States